CLINICAL TRIAL: NCT00704808
Title: Post Marketing Surveillance of Radiotherapy With Concomitant and Adjuvant Chemotherapy With Temozolomide for Patients With Newly Diagnosed and Operated Glioblastoma Multiforme
Brief Title: Post Marketing Surveillance: Newly Diagnosed Glioblastoma Multiforme Treated With Radiotherapy/Temozolomide and Adjuvant Temozolomide (Study P04739)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04739
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Surgical Procedures, Operative; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with newly diagnosed and operated glioblastoma multiforme.
  Interventions: Procedure: Primary surgical treatment; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Procedure: Primary surgical treatment — Primary surgery for tumor resection.
  Other Names: Resection; Operation; Surgery
Radiation: Radiotherapy — Radiotherapy is given with concomitant temozolomide. Dosing according to European Summary of Product Characteristics.
  Other Names: Irradiation; Radiation therapy
Drug: Temozolomide — Temozolomide is first given with concomitant radiotherapy, and then as monotherapy (adjuvant chemotherapy). Dosing according to European Summary of Product Characteristics.
  Other Names: Temodal; Temodar; SCH 052365

SUMMARY:
The purpose of this surveillance is to collect more safety and efficacy data in "non-study" patients during concomitant and adjuvant temozolomide therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed and operated glioblastoma multiforme with postoperative residual tumor <=1.5 cm by magnetic resonance imaging (MRI).
* Age >=18 years.
* Hemoglobin >=10 g/dL.
* White blood cell count >=1.5x10^9/L.
* Platelet count >=100x10^9/L.
* Blood urea <=1.5 x upper limit of normal values (ULN).
* Creatinine <=1.5 x ULN.
* Bilirubin <=1.5 x ULN.
* Aspartate aminotransferase <=3 x ULN.
* Alanine aminotransferase <=3 x ULN.
* Alkaline phosphatase <=2 x ULN.

Exclusion Criteria:

* Tumor-specific pretreatment.
* Contraindication against radiotherapy and/or chemotherapy.
* Malignomas other than basaliomas.
* Existing or planned pregnancy or lactation or inadequate contraception.
* Psychiatric disease.
* Simultaneous participation in another clinical trail or participation in another clinical trail in the last 30 days before recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed glioblastoma multiforme.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Temozolomide: Surgery followed by temozolomide concomitant with radiotherapy (dosed according to the Summary of Product Characteristics [SPC]), then adjuvant monochemotherapy temozolomide (dosed according to the SPC)
Period: Overall Study
Arm/Group | Temozolomide
Started | 180
Completed | 49
Not Completed | 131
Not completed — Discontinued prior to starting treatment | 14
Not completed — Death | 7
Not completed — Tumor progression | 80
Not completed — Patient's decision | 11
Not completed — Early therapy discontinuation | 16
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Treatment change | 1

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age data based on 165 participants (one less than the Intent-to-treat (ITT) population of 166) due to missing data for 1 participant.
  years | 57.65 (11.52)
Sex/Gender, Customized [Number; unit: participants] — Gender information only available for the Intent-to-Treat population of 166 participants.
  participants
    Female | 65
    Male | 101
    Unavailable | 14
Region of Enrollment [Number; unit: participants]
  Germany | 180

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival After Primary Surgical Treatment, Concomitant and Adjuvant Chemotherapy With Temozolomide, for Patients With Newly Diagnosed Glioblastoma Multiforme
Time Frame: After primary surgical treatment and concomitant and adjuvant chemotherapy with temozolomide
Population: Intent-to-Treat population
Measure: Median (Standard Error); unit: Months
Arm/Group | Temozolomide
Number analyzed (Participants) | 166
Months | 9.57 (1.18)

ADVERSE EVENTS:
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 49/166
Other Adverse Events (participants affected / at risk) | 41/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=166)
PANCYTOPENIA (Blood and lymphatic system disorders) | 3 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
PERITONITIS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2)
DEATH (General disorders) | 7 (7)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 7 (8)
IMPAIRED HEALING (General disorders) | 3 (4)
HERPES ZOSTER (Infections and infestations) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
BRAIN OEDEMA (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 4 (4)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 1 (1)
PARTIAL SEIZURES (Nervous system disorders) | 5 (5)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 (5)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1)
SOCIAL STAY HOSPITALISATION (Social circumstances) | 1 (1)
APPENDICECTOMY (Surgical and medical procedures) | 1 (1)
CEREBROSPINAL FLUID DRAINAGE (Surgical and medical procedures) | 1 (1)
CEREBROSPINAL FLUID RESERVOIR PLACEMENT (Surgical and medical procedures) | 1 (1)
HOSPITALISATION (Surgical and medical procedures) | 8 (9)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=166)
CONSTIPATION (Gastrointestinal disorders) | 9 (13)
NAUSEA (Gastrointestinal disorders) | 13 (13)
FATIGUE (General disorders) | 21 (22)
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 (10)
HEADACHE (Nervous system disorders) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publishing or dissemination of study results requires a written approval of the sponsor.